CLINICAL TRIAL: NCT00000840
Title: A Multicenter, Exploratory Study to Evaluate the Effects of Antiretroviral Cessation on Plasma Associated HIV-1 RNA
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: ACTG 304
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-04

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; Zidovudine; Biological Markers; Viremia; RNA, Viral
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Viremia

STUDY DESIGN:
Observational Model: Natural History

SUMMARY:
To evaluate viral load in the blood stream of HIV-infected patients during a 28-day washout following cessation of long-term zidovudine ( AZT ) therapy.

Because viral load (amount of HIV RNA in the plasma) is often used as a measure of the effectiveness of new antiretroviral drugs in clinical trials, a washout period, or cessation of current antiretroviral regimens, is commonly required for study entry to allow for a drug-free steady state of viral load prior to initiation of the new drug. However, the kinetics of the viral rebound following drug withdrawal has not been sufficiently studied, and the proper duration of washout is an estimate.

DETAILED DESCRIPTION:
Because viral load (amount of HIV RNA in the plasma) is often used as a measure of the effectiveness of new antiretroviral drugs in clinical trials, a washout period, or cessation of current antiretroviral regimens, is commonly required for study entry to allow for a drug-free steady state of viral load prior to initiation of the new drug. However, the kinetics of the viral rebound following drug withdrawal has not been sufficiently studied, and the proper duration of washout is an estimate.

Patients who have volunteered to temporarily cease antiretroviral therapy will be followed during a 28-day washout period. Blood samples are drawn at each of nine clinic visits. Patients may resume antiretrovirals after the 28-day washout.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Maintenance therapy for opportunistic infection, provided patient has received at least 1 month of stable therapy prior to study.
* G-CSF.

Patients must have:

* HIV infection.
* CD4 count <= 500 cells/mm3.
* At least 12 months of prior AZT, with 2 months of continuous AZT monotherapy immediately prior to study.
* The need to discontinue AZT because of drug-related toxicity or unwanted side effects or as an entry requirement for another research study.
* Consent of parent or guardian if < 18 years old.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Current medical status that is considered unsuitable for study participation.

Concurrent Medication:

Excluded:

* Therapy for an acute opportunistic infection.

Prior Medication:

Excluded within the past 2 months:

* Antiretrovirals other than AZT.
* Systemic immunomodulators (e.g., gp120, gp160, IL-2, and interferons).

Excluded within the past month:

* Vaccination.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70

CONTACTS AND LOCATIONS:
Overall Officials: Para MF, Study Chair; Demeter L, Study Chair
Locations (8):
- United States (8):
  - Northwestern Univ Med School, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Johns Hopkins Hosp, Baltimore, Maryland
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Case Western Reserve Univ, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Univ of Washington, Seattle, Washington